CLINICAL TRIAL: NCT05724771
Title: Assessing the Safety and Efficacy of Utilizing CGRPmAb Fremanezumab (Ajovy) in Chronic Migraine Patients Currently on Monotherapy OnabotulinumtoxinA (Botox).
Brief Title: COACT Study: CGRPmAbs + OnabotulinumtoxinA Assessment of Chronic Migraine Treatments Study
Acronym: COACT
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chicago Headache Center & Research Institute (Other)
Responsible Party: Principal Investigator, Bradley Torphy, MD, Managing Director, Chicago Headache Center & Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01
Record Dates: First submitted 2023-01-18; First posted 2023-02-13 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Chronic Migraine, Headache
MeSH Terms: conditions — Headache | interventions — fremanezumab

STUDY DESIGN:
Intervention Model Description: Phase IV prospective open label interventional clinical study evaluating beneficial outcomes of the addition of CGRPmAb Fremanezumab in chronic migraine patients currently on monotherapy OnabotulinumtoxinA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Combination of Botox + CGRPmAb (Experimental): OnabotulinumtoxinA + Fremanezumab 225mg/1.5mL = 50
  Interventions: Drug: Combination of Botox + CGRPmAb (Fremanezumab 225mg/1.5mL)

INTERVENTIONS:
Drug: Combination of Botox + CGRPmAb (Fremanezumab 225mg/1.5mL) — OnabotulinumtoxinA + Fremanezumab 225mg/1.5mL

SUMMARY:
Chronic migraine patients treated with OnabotulinumtoxinA may experience breakthrough headaches, especially toward the end of their 12-week therapy. The addition of a CGRPmAb could help in decreasing or eliminating these episodes, but this combination is considered "experimental" by many payers, which often leads to a denial of coverage. Currently, there is no reference in the literature or data to support the treatment of chronic migraine with OnabotulinumtoxinA and CGRPmAbs (Aimovig, Ajovy, Emgality or Vyepti) combination therapy. This has resulted in many patients and providers having to settle for one or the other. Investigators hopes to provide crucial data and findings to support the addition of CGRPmAb in some chronic migraine patients currently on monotherapy OnabotulinumtoxinA.

DETAILED DESCRIPTION:
Phase IV prospective open label interventional clinical study evaluating beneficial outcomes of the addition of CGRPmAb Fremanezumab in chronic migraine patients currently on monotherapy OnabotulinumtoxinA.

The investigators will enroll patients with ≥2 OnabotulinumtoxinA treatments at screening with a history of ≥8 monthly migraine days (average from 3 previous months prior to enrollment (visit 2)). Between visit 1 (screening) and visit 3, all patients will be on monotherapy OnabotulinumtoxinA for up to 12 weeks.

Patients will be administered a total of 2 OnabotulinumtoxinA treatments for the duration of the entire study. OnabotulinumtoxinA treatment will be administered at Day 1 (visit 2) and Day 90 (visit 4), with a treatment window ±6 days.

OnabotulinumtoxinA treatment of 155 units or 195 units will be injected intramuscularly over 31-35 injections of head and neck muscles. Study patients must be on a stable OnabotulinumtoxinA dose at screening (visit 1), that dose will be used for the duration of the study.

Dosing paradigm:

At Day 7 (visit 3) study patients will initiate CGRPmAbs treatment of Fremanezumab 225mg/1.5mL monthly dose for 6 months. Doses will be taken on Days: 7, 37, 67, 97, 127, and 157; with a treatment window ±2 days.

• OnabotulinumtoxinA + Fremanezumab 225mg/1.5mL = 50 Rescue medication will be allowed to treat acute migraine attacks consistent with the parameters referenced in previous CGRP clinical trials.

Acute rescue utilizing -gepants will be limited to no more than 5 days per month.

No use of -gepants as a preventative treatment for at least 1 week prior to screening (visit 1) and throughout the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic migraine patients between 18 to 75 years old
* Chronic migraine patients with ≥ 12-month history of migraine
* Participant has received at least 2 consecutive OnabotulinumtoxinA treatment at screening (visit 1)
* Achieved a clinically appropriate response from monotherapy OnabotulinumtoxinA at enrollment (visit 2):

  * ≥50% reduction in mean monthly headache days of at least moderate severity OR Reduction of ≥7 mean monthly headache days of at least moderate severity OR
  * HIT-6 reduction of ≥5 points
* History of ≥8 monthly migraine days (average from 3 previous months prior to enrollment (visit 2))

Exclusion Criteria:

* History of <8 monthly migraine days (average from 3 previous months prior to enrollment (visit 2))
* Patients with current use, or use within 3 months prior to screening (visit 1) a CGRPmAbs (Aimovig, Ajovy, Emgality, or Vyepti)
* Concomitant use of gepants as a preventative treatment < 1 week prior to screening (visit 1).
* Utilizing gepants as an acute rescue treatment >5 days per month.
* Current user of recreational or illicit drugs, or a history within 1 year prior to screening (visit 1) of drug or alcohol abuse or dependence
* Clinically significant hematologic, endocrine, cardiovascular, pulmonary, gastrointestinal, or neurologic disease. If there is a history of such a disease, but the condition has been stable for more than 1 year prior to screening (visit 1) and is judged by the PI as not likely to interfere with participation in the study, the participant may be included.
* Female is pregnant, planning to become pregnant during the course of the study, or currently lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change in number of monthly migraine days with the addition of CGRPmAb Fremanezumab in chronic migraine patients currently on monotherapy OnabotulinumtoxinA. | 6 months
  Change in number of monthly migraine days from baseline.

SECONDARY OUTCOMES:
To assess improvements in HIT-6 (Headache Impact Test) score of >5 point reduction with the addition of CGRPmAb Fremanezumab in chronic migraine patients currently on monotherapy OnabotulinumtoxinA. | 6 months
  Change in HIT-6 (Headache Impact Test) assessment score from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Chicago Headache Center & Research Institute, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goadsby PJ, Reuter U, Hallstrom Y, Broessner G, Bonner JH, Zhang F, Sapra S, Picard H, Mikol DD, Lenz RA. A Controlled Trial of Erenumab for Episodic Migraine. N Engl J Med. 2017 Nov 30;377(22):2123-2132. doi: 10.1056/NEJMoa1705848. PMID 29171821
- [Background] Dodick DW, Ashina M, Brandes JL, Kudrow D, Lanteri-Minet M, Osipova V, Palmer K, Picard H, Mikol DD, Lenz RA. ARISE: A Phase 3 randomized trial of erenumab for episodic migraine. Cephalalgia. 2018 May;38(6):1026-1037. doi: 10.1177/0333102418759786. Epub 2018 Feb 22. PMID 29471679
- [Background] Stauffer VL, Dodick DW, Zhang Q, Carter JN, Ailani J, Conley RR. Evaluation of Galcanezumab for the Prevention of Episodic Migraine: The EVOLVE-1 Randomized Clinical Trial. JAMA Neurol. 2018 Sep 1;75(9):1080-1088. doi: 10.1001/jamaneurol.2018.1212. PMID 29813147
- [Background] Skljarevski V, Matharu M, Millen BA, Ossipov MH, Kim BK, Yang JY. Efficacy and safety of galcanezumab for the prevention of episodic migraine: Results of the EVOLVE-2 Phase 3 randomized controlled clinical trial. Cephalalgia. 2018 Jul;38(8):1442-1454. doi: 10.1177/0333102418779543. Epub 2018 May 31. PMID 29848108
- [Background] Dodick DW, Silberstein SD, Bigal ME, Yeung PP, Goadsby PJ, Blankenbiller T, Grozinski-Wolff M, Yang R, Ma Y, Aycardi E. Effect of Fremanezumab Compared With Placebo for Prevention of Episodic Migraine: A Randomized Clinical Trial. JAMA. 2018 May 15;319(19):1999-2008. doi: 10.1001/jama.2018.4853. PMID 29800211
- [Background] Ferrari MD, Diener HC, Ning X, Galic M, Cohen JM, Yang R, Mueller M, Ahn AH, Schwartz YC, Grozinski-Wolff M, Janka L, Ashina M. Fremanezumab versus placebo for migraine prevention in patients with documented failure to up to four migraine preventive medication classes (FOCUS): a randomised, double-blind, placebo-controlled, phase 3b trial. Lancet. 2019 Sep 21;394(10203):1030-1040. doi: 10.1016/S0140-6736(19)31946-4. Epub 2019 Aug 16. PMID 31427046
- [Background] Blumenfeld AM, Frishberg BM, Schim JD, Iannone A, Schneider G, Yedigarova L, Manack Adams A. Real-World Evidence for Control of Chronic Migraine Patients Receiving CGRP Monoclonal Antibody Therapy Added to OnabotulinumtoxinA: A Retrospective Chart Review. Pain Ther. 2021 Dec;10(2):809-826. doi: 10.1007/s40122-021-00264-x. Epub 2021 Apr 21. PMID 33880725